CLINICAL TRIAL: NCT06215209
Title: Physiological Effect of Prone Position in Patients With Ultra-low Tidal Volume Ventilation
Brief Title: Effect of PP in Patients With Ultra-low VT
Status: Recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Director of Intensive Care Unit, Principal Investigator, Clinical Professor, Southeast University, China
Other Study IDs: Ultra-low VT and PP
Record Dates: First submitted 2024-01-10; First posted 2024-01-22 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Acute Respiratory Distress Syndrome; Prone Position; Tidal Volume
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Patient Positioning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultra-low tidal volume group: ARDS patients with ultra-low tidal volume ventilation
  Interventions: Other: position

INTERVENTIONS:
Other: position — patients will be in supine position and prone position

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a heterogeneous syndrome with similar clinicopathological feathers caused by different etiologies. Respiratory supportive strategies is the main ARDS management, and the guidelines recommend low tidal volume to improve clinical outcomes. To be note, overdistension can still occur even if using a tidal volume as low as 6 ml/kg, given the heterogeneous nature of the syndrome. Therefore, adjusting tidal volume level to less than 6ml/kg may reduce ventilator-induced lung injury (VILI) and thus improve outcomes, especially in patients with severe lung injury. Prone position is also an important management in severe ARDS. Prone position can improve ventilation-perfusion (V/Q) matching and reduce the risk of VILI by recruiting dorsal collapsed alveoli. Meanwhile, prone position has also been shown to improve hemodynamics. Recent studies have showed that prone position did not reduce duration of venovenous extracorporeal membrane oxygenation (VV-ECMO) and 90-day mortality in patients with ARDS who receive VV-ECMO with ultra-low tidal volume ventilation. Therefore, the effect of PP on ventilation and lung blood flow in ARDS patients treated with VV-ECMO wiht ultra-low tidal volume ventilation remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients were enrolled if they were undergoing invasive mechanical ventilation and were supported by VV-ECMO for less than 48 hours

Exclusion Criteria:

* younger than 18 years old
* contraindications for prone position ventilation
* past chronic respiratory diseases (long-term family oxygen therapy for chronic
* respiratory diseases such as pulmonary fibrosis or COPD)
* New York Heart Association class above II
* contraindications to the use of EIT (e.g., presence of pacemaker or chest surgical wounds dressing) or prone position (as decided by the attending physician)
* severe hemodynamic instability
* gave written or witnessed verbal informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ARDS admitted to the Department of Critical Care Medicine, Zhongda Hospital, Southeast University and receiving VV-ECMO treatment
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
ventilation-perfusion mathching | up to 24 hours
  ventilation-perfusion matching will be monitored using an EIT monitor (PulmoVista® 500, Dräger, Lübeck, Germany) in supine position and prone position

SECONDARY OUTCOMES:
The percentage of shunt | up to 24 hours
  The percentage of shunt will be monitored using an EIT monitor (PulmoVista® 500, Dräger, Lübeck, Germany) in supine position and prone position
The percentage of dead space | up to 24 hours
  The percentage of shunt will be monitored using an EIT monitor (PulmoVista® 500, Dräger, Lübeck, Germany) in supine position and prone position
The percentage of dorsal ventilation | up to 24 hours
  The percentage of dorsal ventilation will be monitored using an EIT monitor (PulmoVista® 500, Dräger, Lübeck, Germany) in supine position and prone position
The percentage of dorsal perfusion | up to 24 hours
  The percentage of dorsal ventilation will be monitored using an EIT monitor (PulmoVista® 500, Dräger, Lübeck, Germany) in supine position and prone position
Center of ventilation (CoV) | up to 24 hours
  Center of ventilation will be monitored using an EIT monitor (PulmoVista® 500, Dräger, Lübeck, Germany) in supine position and prone position
Regional ventilation delay (RVD) | up to 24 hours
  Regional ventilation delay will be monitored using an EIT monitor (PulmoVista® 500, Dräger, Lübeck, Germany) in supine position and prone position
Arterial blood gas analysis | up to 24 hours
  Arterial blood gas analysis included pH, PaO2, PaCO2 and PaO2/FiO2 in supine position and prone position
Respiratory system compliance | up to 24 hours
  Respiratory system compliance will be monitored in supine position and prone position.

CONTACTS AND LOCATIONS:
Overall Officials: liu ling, phD, Study Chair — Zhongda Hospital
Locations (1):
- Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China